CLINICAL TRIAL: NCT01827449
Title: Hypothermia Rewarming Effectiveness of Distal Limb Warming With Either Fluidotherapy or Warm Water Immersion
Brief Title: Hypothermia Rewarming With Distal Limb Warming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr.Gordon Giesbrecht, Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2013:039; NSERC 2011-6 (Other Grant/Funding Number: NSERC Discovery Grant)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Rewarming by Shivering Heat Production Only; Rewarming by Arm and Leg Immersion in Warm Water; Rewarming by Arm and Leg Exposure to Fluidotherapy
Keywords: rewarming; core cooling; afterdrop; hospital treatment; hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fluidotherapy warming device — Device uses airborne heated cellulose particles which are blown against the skin to provide convective warming.
  Other Names: Chattanooga Fluidotherapy model 115D

SUMMARY:
The study will compare the rewarming effectiveness of heat donation through the distal arms and legs during rewarming of mildly hypothermic subjects. Warming will be accomplished through either warm water immersion; and fluidotherapy. The investigators hypothesize that fluidotherapy will be as, or more, effective compared to warm water immersion

DETAILED DESCRIPTION:
Dr. Gordon Giesbrecht is studying/comparing the effectiveness of heat donation through the distal arms and legs in rewarming a mildly hypothermic individual. Warming will be accomplished through either warm water immersion; and fluidotherapy.

Procedure. Eight participants will be cooled in 8°C water on three occasions and then warmed by each of three warming conditions. The study will include following specific procedures: Anthropometric data which includes age, weight, height, and measurements of skinfold thickness at four sites- biceps, triceps, subscapularis, and suprailiac will be collected. Participant's heart rate and electrocardiogram will be monitored continuously throughout the experiment.

Participants will be instrumented as follows:

1. About 12 heat flux disks (2 cm in diameter) will be taped to the skin on the arms, legs, torso, head etc. to measure skin temperature and heat transfer from the skin.
2. Three ECG leads will be affixed to the skin.
3. Core temperature will be measured with a disposable esophageal thermocouple. A thin, flexible tube will be inserted through the nose, to midway down the esophagus at the level of the heart.
4. Oxygen consumption will be continuously measured with a metabolic cart. Participants will be asked to wear a face mask which will collect the expired breath during the cooling as well as the rewarming periods.

Conditions: The three treatment methods are as follows.

A. Spontaneous rewarming (Shivering only) - In this control condition, no external heat will be provided and the participant will rewarm spontaneously with the heat produced from shivering.

B. Warm water distal extremities immersion - Distal arms and legs will be immersed in warm water at 45°C for rewarming.

C.Fluidotherapy distal extremities rewarming - Distal arms and legs will be immersed in Fluidotherapy equipment for rewarming at 50°C.

Rewarming procedures will be administered either for a period of 60 minutes or until core temperature returns to normal values ( ̴ 36.5-37˚C). Following that, participants will be placed in a warm water bath (40-42˚C).

Research Design: Each of the three experimental trials, separated by at least 48 hours. On each of the three trials, participants will be immersed up to the level of the sternal notch in 8˚C for up to 60 minutes or until the core temperature falls to 35˚C. The participant will then exit the water, be dried off and rewarmed with either lie inside a vapor barrier within a hooded sleeping bag with the head inside the hood, or sitting with their distal arms and legs immersed in either Fluidotherapy at 50°C or warm water at 45°C. The rewarming will be administered for 60 minutes or until the core temperature returns to normal values (̴36.5-37˚C). The order of warming methods will follow a balanced design.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 yrs old, males or females, healthy

Exclusion Criteria:

* cardiopulmonary disease
* any symptoms caused by cold exposure

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Core temperature rewarming rate | Sixty minutes post-cooling
  Esophageal temperature will be measured to determine the rate of core temperature increase during rewarming periods

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada